CLINICAL TRIAL: NCT01993238
Title: An Evaluation of Procedural Analgesia for Out-Patient Liposonix Treatment
Brief Title: Evaluation of Procedural Analgesia for Liposonix Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solta Medical (Industry)
Responsible Party: Sponsor
Organization: Valeant Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-140-LP-H
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Body Contouring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposonix with pre-treatment analgesia (Experimental): Liposonix System (Model 2) treatment of subcutaneous adipose tissue with pre-treatment analgesia (combination of ondansetron, ketorolac, and hydromorphone)
  Interventions: Device: Liposonix System (Model 2); Drug: Pre-treatment analgesia

INTERVENTIONS:
Device: Liposonix System (Model 2) — Treatment of subcutaneous adipose tissue of the abdomen using high intensity focused ultrasound (Liposonix System Model 2).
Drug: Pre-treatment analgesia — Pre-treatment analgesia (combination of ondansetron, ketorolac, and hydromorphone)

SUMMARY:
The objectives of this study are to evaluate the safety and effectiveness of procedural analgesia for improvements in tolerability of treatment with the Liposonix System.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult female or male, 18 to 65 years of age.
* Subject must weigh more than 120 pounds.
* Subject must have a Body Mass Index of ≤ 30 kg/m2.
* Subject must have thickness of skin + subcutaneous adipose tissue in the anticipated treatment area of ≥ 2.3 cm.
* Subject must be able to read, write, speak, and understand English.

Exclusion Criteria:

* Female subject who is pregnant, is suspected to be pregnant, or is lactating
* Subjects diagnosed with coagulation disorders or are receiving anticoagulant therapy or medications or dietary supplements which impede coagulation or platelet aggregation
* Subject has diabetes or cardiovascular disease
* Subject has had any aesthetic procedure to the region to be treated within past 6 months
* Subject has systemic skin disease or skin disease in the area to be treated
* Subject has any abnormality of the skin or soft tissues of the abdominal wall in the area to be treated
* Subject has had previous open or laparoscopic surgery in the anticipated treatment area
* Subjects is on prescription or over the counter weight reduction medication or programs, or had weight reduction procedures
* Subject has skin or superficial tissue that does not lie flat on its own when the subject is in the supine position
* Subjects undergoing chronic steroid or immunosuppressive therapy
* Subjects who have cardiac pacemakers or any implantable electrical device
* Subjects who have metal implants of any type in the area to be treated
* History of cancer
* Subjects who have sensory loss or dysesthesia in the area to be treated
* Subjects taking chronic benzodiazepines or opiates
* Subjects with a history of severe nausea/vomiting with opioid analgesics
* Subjects with sleep apnea
* Subjects with known allergies or sensitivities to study drugs
* Subjects with liver disease
* Subjects with renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wheeland, MD, Principal Investigator; Reid Rubsamen, MD, Principal Investigator
Locations (1):
- Solta Medical Aesthetic Center, Hayward, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposonix With Pre-treatment Analgesia
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Arm/Group | Liposonix With Pre-treatment Analgesia
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain Score for Overall Treatment
Description: Following treatment, the subject was asked to evaluate the pain level for the overall treatment using the 0-10 Visual Analog Scale (0 represents no pain and 10 represents worst imaginable pain)
Time Frame: Baseline
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposonix With Pre-treatment Analgesia
Number analyzed (Participants) | 11
units on a scale | 6.3 (2.2)

2. Secondary Outcome: Safety Assessment
Description: Adverse events will be assessed and documented throughout the study
Time Frame: Baseline, 1 day, 1 week
Reporting Status: Not Posted

3. Secondary Outcome: Pain Scores Reported at 1-day Post-Treatment
Description: During the 1-day follow-up phone call, subjects were asked to rate the pain they were currently experiencing from the Liposonix treatment using a 0-10 pain scale (0 represents no pain and 10 represents worst pain imaginable).
Time Frame: 1 day
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposonix With Pre-treatment Analgesia
Number analyzed (Participants) | 11
units on a scale | 2.1 (2.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from day 0 through study follow-up (1 week post-treatment)
Arm/Group | Liposonix With Pre-treatment Analgesia
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposonix With Pre-treatment Analgesia (N=11)
Car Accident (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient admitted to hospital following car accident for lower back pain. Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposonix With Pre-treatment Analgesia (N=11)
Pain during treatment (General disorders) | 11 (11)
Ecchymosis (Skin and subcutaneous tissue disorders) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 11 (11)
Tenderness (Skin and subcutaneous tissue disorders) | 5 (5)
Soreness (Skin and subcutaneous tissue disorders) | 5 (5)
Tingling/Altered Sensation (Skin and subcutaneous tissue disorders) | 5 (5)
Edema (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea/Vomiting (General disorders) | 3 (3)
Dizziness/Feeling Faint (General disorders) | 2 (2)
Warm sensation on treatment area (Skin and subcutaneous tissue disorders) | 2 (2)
Surface sensitivity/soreness at treatment site (Skin and subcutaneous tissue disorders) | 2 (2)
Tiredness (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Bruising at attempted IV site (Skin and subcutaneous tissue disorders) | 1 (1)
Burning sensation to touch (Skin and subcutaneous tissue disorders) | 1 (1)
Pain with movement (General disorders) | 1 (1)
Sense of pressure at treatment site (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall notify Sponsor of the intent to publish or present independent Study Data, and agrees not to publish or publicly present and/or discuss such data, Investigator's current findings and/or the results of the Study independently without the express written consent of Sponsor, which consent may be withheld. Prior to submission for publication or presentation, all draft manuscripts must be submitted, reviewed and approved by Sponsor for confidential material.